CLINICAL TRIAL: NCT05075720
Title: Randomised Controlled Trial to Investigate N-nitrosamine Formation After Meat Intake - Meat Study of the Nitrate INFORMER Studies; Nitrate INFORMER Studies: Is Nitrosamine FORMation dEpenent on souRce
Brief Title: Nitrate INFORMER Meat Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edith Cowan University (Other)
Collaborators: The University of Western Australia (Other); Flinders University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-02629-BONDONNO
Record Dates: First submitted 2021-08-30; First posted 2021-10-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Health Risk Behaviors
MeSH Terms: conditions — Health Risk Behaviors | interventions — Meat

STUDY DESIGN:
Intervention Model Description: prospective, mono-centre, randomised, controlled, crossover study
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the interventions, participants, and the investigators responsible for delivering the interventions will be unblinded throughout the trial. However, all researchers performing the laboratory analyses and data analyses will be blinded to the interventions that the participants received until after the data analysis has been performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Supplement: Meat with added nitrate (Experimental): The intervention comprises 50 g salami and 35 g ham on white bread sandwich at breakfast and lunch.
  This intervention will allow us to determine both endogenous formation of N-nitrosamines as well as N-nitrosamines present in the commercially prepared meat.
  Interventions: Dietary Supplement: Meat without added nitrate; Dietary Supplement: Control
- Dietary Supplement: Meat without added nitrate (Experimental): The intervention comprises 65 g Pork mince on white bread sandwich at breakfast and lunch. Nitrate is not an allowed additive in pork mince.
  This intervention will allow us to determine if there is endogenous formation of N-nitrosamines as well as N-nitrosamines present in the prepared meat due to the natural content of nitrate in meat.
  Interventions: Dietary Supplement: Meat with added nitrate; Dietary Supplement: Control
- Dietary Supplement: Control (Sham Comparator): The control comprises low nitrate vegetable protein burger on white bread. Protein content matched to interventions 1 and 2.
  Interventions: Dietary Supplement: Meat with added nitrate; Dietary Supplement: Meat without added nitrate

INTERVENTIONS:
Dietary Supplement: Meat with added nitrate — The intervention comprises 50 g salami and 35 g ham on white bread sandwich at breakfast and lunch.
  This intervention will allow us to determine both endogenous formation of N-nitrosamines as well as N-nitrosamines present in the commercially prepared meat.
  Arms: Dietary Supplement: Control; Dietary Supplement: Meat without added nitrate
Dietary Supplement: Meat without added nitrate — The intervention comprises 65 g Pork mince on white bread sandwich at breakfast and lunch. Nitrate is not an allowed additive in pork mince.
  This intervention will allow us to determine if there is endogenous formation of N-nitrosamines as well as N-nitrosamines present in the prepared meat due to the natural content of nitrate in meat.
  Arms: Dietary Supplement: Control; Dietary Supplement: Meat with added nitrate
Dietary Supplement: Control — The control comprises low nitrate vegetable protein burger on white bread. Protein content matched to interventions 1 and 2.
  Arms: Dietary Supplement: Meat with added nitrate; Dietary Supplement: Meat without added nitrate

SUMMARY:
Nitrate is a controversial component of vegetables, meat, and drinking water. The now well-established benefits of nitrate, through the enterosalivary nitrate-nitrite-nitric oxide (NO) pathway, on cardiovascular risk factors and long-term cardiovascular disease risk are tarnished by a continuing concern about a link between nitrate ingestion and cancer. This can result in misguided advice to avoid consumption of high-nitrate leafy green vegetables by both the media and the scientific literature. A recent media headline stated, "Cancer alert over rocket: trendy salad leaves exceed safe levels of carcinogenic nitrates in one in every ten samples". One scientific review stated, "the presence of nitrate in vegetables, as in water and generally in other foods, is a serious threat to man's health". Controversy in the literature, and gaps in the knowledge are leading to confusing messages around vegetables that may play a critical role in cardiovascular health.

The major dietary sources of nitrate are vegetables, meat, and drinking water. Source of nitrate could be a crucial factor determining whether the consumption of nitrate is linked with beneficial (such as improving cardiovascular health) versus harmful (N-nitrosamine formation) effects. For example, unlike meat and water-derived nitrate, vegetables contain high levels of vitamin C and/or polyphenols that may inhibit the production of N-nitrosamines. So far, no study has investigated the formation of N-nitrosamines after consumption of these different sources in humans. This study will compare N-nitrosamine formation after intake of meat with and without added nitrate.

DETAILED DESCRIPTION:
Study design

A crossover study design will be used with a 1-week washout period between interventions. Participants diet for the day before and the day of the intervention will be standardised (food choices on visit 1 will be matched for visit 2) as follows:

For the day before the study visit:

* A choice of 3 breakfasts: cornflakes with milk; rice krispies with milk; white bread toast with eggs.
* Lunch will be provided comprising pumpkin soup and white bread/or rice
* Dinner: a low nitrate vegetarian meal
* All water will be provided
* Participants will be asked to refrain from drinking coffee and any alcoholic beverage and do any exercise 24 hours prior to their study visit.

For the day of the study visit:

* Participants will arrive at the study unit fasting
* Breakfast and lunch will comprise the intervention
* Participants will be provided with a standardised dinner: a low nitrate vegetarian meal
* All water will be provided
* Participants will be asked to refrain from drinking coffee and any alcoholic beverage and do any exercise for 24 hours from the time of the first intervention.

Dietary interventions

1. Meat with added nitrate: 50 g salami and 35 g ham on white bread sandwich at breakfast and lunch.

   This intervention will allow us to determine both endogenous formation of N-nitrosamines as well as N-nitrosamines present in the commercially prepared meat.
2. Meat without added nitrate: 65 g Pork mince on white bread sandwich at breakfast and lunch. Nitrate is not an allowed additive in pork mince.

   This intervention will allow us to determine if there is endogenous formation of N-nitrosamines as well as N-nitrosamines present in the prepared meat due to the natural content of nitrate in meat.
3. Control: low nitrate vegetable protein burger on white bread. Protein content matched to interventions 1 and 2.

Allocation Sequence generation. The sequence of intervention allocation will be generated via block randomisation using computer-generated random numbers. Random block sizes of 2 and 4 will be used.

Concealment mechanism. Fifty randomly generated sequences of the interventions for each of the study participants will be printed on separate pieces of paper and sealed in opaque envelopes, numbered 1-50, by a study investigator not involved in performing the intervention, the data collection or the data analysis.

Implementation. Once a participant is deemed eligible and enrolled in the study, the study coordinator will contact the study investigator responsible for randomisation and intervention allocation to obtain the next available envelope and randomly generated intervention sequence.

Blinding Given the nature of the interventions, participants, and the investigators responsible for delivering the interventions will be unblinded throughout the trial. However, all researchers performing the laboratory analyses and data analyses will be blinded to the interventions that the participants received until after the data analysis has been performed.

Participant timeline Prior to the first clinic visit, each participant will complete a food frequency questionnaire (FFQ) to assess background habitual diet.

At each clinic visit, a baseline urine and faecal stool sample will be collected for measurement of N-nitrosamines. Prior to the intervention participants will be instructed to void their bladder into baseline urine collection container. After the first intervention all urine for the subsequent 24-hour period will be collected for measurement of N-nitrosamines, nitrate, and nitrite. A faecal stool will be collected for measurement of N-nitrosamines, nitrate, and nitrite.

Assessments

Urine and faecal stool collection. A urine sample will be collected at baseline, and from intervention up until 24 hours post-intervention. For the baseline sample, participants will be provided with a sterilized container and instructions to discard the first urine sample of the day and then collect all urine until the intervention which will be brought into the clinic. Participants will be instructed to drink 250 ml water on waking. For the 24-hour urine samples, participants will be provided with sterilized containers and instructions to collect all urine until 24 hours post intervention. Urine aliquots will be frozen at -80°C until analysis. A stool sample will be collected at baseline and for the 24 hour period post the first intervention. Participants will be provided with instructions and a stool sample collection pack (collection bags, cable ties, large zip lock bags, freezer ice blocks and a designated cooler bag for transport). Collected stool samples will be weighed and frozen at -80°C until analysis.

N-nitrosamines. Nitrosamines in the interventions, urine and stool samples will be measured by gas chromatography mass spectrometry (GCMS). Volatile nitrosamines will be extracted with dichloromethane and are well separated by gas chromatography. Identification will be by retention time and unique molecular ions for each of five common nitrosamines. Quantitation will be made by using deuterium labelled internal standards, N-nirtrosodimethylamine-D6; N-nitrosodiethylamine D10; N-nitrosomorpholine D8 (Cambridge Isotopes) and N-nitrosopiperidine D10 (Toronto Research Chemicals). The most commonly detected nitrosamines are NDMA and N-Nitrosopiperidine (NPIP). Control experiments in which water stored in the same containers as those used for sample collection and storage will be performed to test for any leaching of volatile nitrosamines.

Sample size and power

Sample size is based on a crossover design and the primary outcome of N-nitrosamines, specifically N-Nitrosodimethylamine (NDMA) in urine. At α=0.05, 2 measures per subject (baseline and post) and a correlation of ρ=0.6 between measures, 25 participants will provide 80% power to detect a 0.6 SD increase in NDMA concentration. To allow for a 10% withdrawal rate, we plan to recruit 25 participants into the study. A rolling recruitment of participants will be performed until the sample size is reached.

Statistical methods

Statistical analyses will be performed using IBM SPSS Statistics for Windows, version 25 (IBM) and STATA/IC 17.0 (StataCorp LLC). Descriptive statistics of normally distributed continuous variables will be expressed as mean (± standard deviation, SD), non-normally distributed continuous variables as median (interquartile range, IQR) and categorical variables as number (proportion, %). Data will be assessed for outliers and normality prior to analysis. Non-normally distributed data will be log transformed if necessary. Treatment effects for outcomes will be obtained using linear mixed models including baseline measurements, treatment order, period, and time (as a categorical variable) as fixed effects. We will also include a treatment X period interaction term to assess for possible treatment-period interactions and we will separately assess for carryover effects with dummy variables to indicate the previous treatment. Treatment effects for outcomes with a single post-intervention measurement will be obtained using linear mixed models including baseline measurements, treatment order, and period as predictors. The subject ID number will be included as a random intercept in each model. An overall 2-sided type-1 error rate of P<0.05 will be used to assess statistical significance for all hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

The recruitment will be as inclusive as possible so that the results are relevant to much of the general population. Twenty-five men and women will be recruited from the Perth general population according to the following criteria:

* aged between 18 to 70 years old
* healthy, ambulant, community-dwelling
* with no history of major chronic disease

Exclusion Criteria:

Individuals volunteering to participate in the study will be excluded according to the following criteria:

* current or recent (<12 months) smoking
* body mass index (BMI) <18 or > 35 kg/m2
* systolic blood pressure > 160 mmHg
* diastolic blood pressure > 100 mmHg
* any major illness such as cancer, psychiatric illness, diagnosed diabetes
* use of any of the following medications: statins, antihypertensives, nitric oxide donors, antithrombotic medication, anti-coagulant medication, anti-arrhythmic drugs, beta-blockers, regular aspirin use, regular proton pump inhibitor use
* alcohol consumption > 30g/day
* who are pregnant, lactating, or wishing to become pregnant during the study
* use of antibiotics within the previous 12 weeks of the study
* regular use of mouthwash and not willing to cease mouthwash use for the duration of the study
* participation on other research studies
* major gastrointestinal tract condition e.g. Crohns disease and inflammatory bowel disease
* and inability or unwillingness to follow the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
N-nitrosamines in urine post intervention (up to 24 hours) | At each clinic visit, all urine from the start of intervention up till 24 hours will be collected.
  Participants will be provided with sterilized containers and instructions to collect all urine until 24 hours post intervention. Urine aliquots will be frozen at -80°C until analysis. N-nitrosamines will be measured by gas chromatography mass spectrometry (GCMS).
N-nitrosamines in stool samples post intervention (up to 24 hours) | At each clinic visit, all stool samples from the start of intervention up till 24 hours will be collected.
  Participants will be provided with instructions and a stool sample collection pack (collection bags, cable ties, large zip lock bags, freezer ice blocks and a designated cooler bag for transport). Collected stool samples will be weighed and frozen at -80°C until analysis. N-nitrosamines will be measured by gas chromatography mass spectrometry (GCMS).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine P Bondonno, PhD, RNutr., Principal Investigator — Edith Cowan University
Locations (1):
- Royal Perth Hospital Research Foundation, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lundberg JO, Weitzberg E. NO-synthase independent NO generation in mammals. Biochem Biophys Res Commun. 2010 May 21;396(1):39-45. doi: 10.1016/j.bbrc.2010.02.136. PMID 20494108
- [Result] Blekkenhorst LC, Bondonno NP, Liu AH, Ward NC, Prince RL, Lewis JR, Devine A, Croft KD, Hodgson JM, Bondonno CP. Nitrate, the oral microbiome, and cardiovascular health: a systematic literature review of human and animal studies. Am J Clin Nutr. 2018 Apr 1;107(4):504-522. doi: 10.1093/ajcn/nqx046. PMID 29635489
- [Result] Bondonno CP, Blekkenhorst LC, Liu AH, Bondonno NP, Ward NC, Croft KD, Hodgson JM. Vegetable-derived bioactive nitrate and cardiovascular health. Mol Aspects Med. 2018 Jun;61:83-91. doi: 10.1016/j.mam.2017.08.001. Epub 2017 Sep 7. PMID 28802834
- [Result] Spiegelhalder B, Eisenbrand G, Preussmann R. Influence of dietary nitrate on nitrite content of human saliva: possible relevance to in vivo formation of N-nitroso compounds. Food Cosmet Toxicol. 1976 Dec;14(6):545-8. doi: 10.1016/s0015-6264(76)80005-3. No abstract available. PMID 1017769
- [Result] Tannenbaum SR, Weisman M, Fett D. The effect of nitrate intake on nitrite formation in human saliva. Food Cosmet Toxicol. 1976 Dec;14(6):549-52. doi: 10.1016/s0015-6264(76)80006-5. No abstract available. PMID 1017770
- [Result] Gangolli SD, van den Brandt PA, Feron VJ, Janzowsky C, Koeman JH, Speijers GJ, Spiegelhalder B, Walker R, Wisnok JS. Nitrate, nitrite and N-nitroso compounds. Eur J Pharmacol. 1994 Nov 1;292(1):1-38. doi: 10.1016/0926-6917(94)90022-1. PMID 7867685
- [Result] Mirvish SS. Role of N-nitroso compounds (NOC) and N-nitrosation in etiology of gastric, esophageal, nasopharyngeal and bladder cancer and contribution to cancer of known exposures to NOC. Cancer Lett. 1995 Jun 29;93(1):17-48. doi: 10.1016/0304-3835(95)03786-V. PMID 7600541
- [Result] IARC Working Group on the Evaluation of Carcinogenic Risks to Humans. IARC monographs on the evaluation of carcinogenic risks to humans. Ingested nitrate and nitrite, and cyanobacterial peptide toxins. IARC Monogr Eval Carcinog Risks Hum. 2010;94:v-vii, 1-412. No abstract available. PMID 21141240
- [Result] Hord NG, Tang Y, Bryan NS. Food sources of nitrates and nitrites: the physiologic context for potential health benefits. Am J Clin Nutr. 2009 Jul;90(1):1-10. doi: 10.3945/ajcn.2008.27131. Epub 2009 May 13. PMID 19439460
- [Result] Blekkenhorst LC, Prince RL, Ward NC, Croft KD, Lewis JR, Devine A, Shinde S, Woodman RJ, Hodgson JM, Bondonno CP. Development of a reference database for assessing dietary nitrate in vegetables. Mol Nutr Food Res. 2017 Aug;61(8). doi: 10.1002/mnfr.201600982. Epub 2017 May 3. PMID 28105786
- [Result] Bartsch H, Ohshima H, Pignatelli B. Inhibitors of endogenous nitrosation. Mechanisms and implications in human cancer prevention. Mutat Res. 1988 Dec;202(2):307-24. doi: 10.1016/0027-5107(88)90194-7. PMID 3057363
- [Result] Levallois P, Ayotte P, Van Maanen JM, Desrosiers T, Gingras S, Dallinga JW, Vermeer IT, Zee J, Poirier G. Excretion of volatile nitrosamines in a rural population in relation to food and drinking water consumption. Food Chem Toxicol. 2000 Nov;38(11):1013-9. doi: 10.1016/s0278-6915(00)00089-2. PMID 11038239
- [Result] Bartholomew B, Hill MJ. The pharmacology of dietary nitrate and the origin of urinary nitrate. Food Chem Toxicol. 1984 Oct;22(10):789-95. doi: 10.1016/0278-6915(84)90116-9. PMID 6541617
- [Result] Bondonno CP, Croft KD, Puddey IB, Considine MJ, Yang X, Ward NC, Hodgson JM. Nitrate causes a dose-dependent augmentation of nitric oxide status in healthy women. Food Funct. 2012 May;3(5):522-7. doi: 10.1039/c2fo10206d. Epub 2012 Feb 16. PMID 22336776
- [Result] Bondonno CP, Downey LA, Croft KD, Scholey A, Stough C, Yang X, Considine MJ, Ward NC, Puddey IB, Swinny E, Mubarak A, Hodgson JM. The acute effect of flavonoid-rich apples and nitrate-rich spinach on cognitive performance and mood in healthy men and women. Food Funct. 2014 May;5(5):849-58. doi: 10.1039/c3fo60590f. PMID 24676365
- [Result] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Result] Cole JR, Wang Q, Fish JA, Chai B, McGarrell DM, Sun Y, Brown CT, Porras-Alfaro A, Kuske CR, Tiedje JM. Ribosomal Database Project: data and tools for high throughput rRNA analysis. Nucleic Acids Res. 2014 Jan;42(Database issue):D633-42. doi: 10.1093/nar/gkt1244. Epub 2013 Nov 27. PMID 24288368
- [Result] Parks DH, Chuvochina M, Waite DW, Rinke C, Skarshewski A, Chaumeil PA, Hugenholtz P. A standardized bacterial taxonomy based on genome phylogeny substantially revises the tree of life. Nat Biotechnol. 2018 Nov;36(10):996-1004. doi: 10.1038/nbt.4229. Epub 2018 Aug 27. PMID 30148503

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT05075720/Prot_SAP_000.pdf